CLINICAL TRIAL: NCT05973864
Title: A Phase II Study to Evaluate CAPecitabine Plus Pembrolizumab as Post-operative Adjuvant Therapy for Triple Negative Breast Cancer With Residual Disease After Neoadjuvant Chemo-immunotherapy
Brief Title: Capecitabine Plus Pembrolizumab in Patients With Triple Negative Breast Cancer After Chemo-immunotherapy and Surgery
Acronym: CAPPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2211; 2023-505291-30-01 (Other: EU CT number)
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Triple Negative Breast Neoplasms
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pembrolizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm : Pembrolizumab and capecitabine (Experimental): * Pembrolizumab will be administered at a fixed dose of 200 mg every 3 weeks (Q3W), with a total of 9 cycles at adjuvant phase of the treatment;
  * Capecitabine will be administrated at a dose of 1250 mg/m² twice a day (BID) (14 days on / 7 days off) for a total of 8 cycles, with a dose reduction at 825 mg/m² BID during radiotherapy if indicated
  * Local radiotherapy will be performed as per standard practice if indicated.
  Interventions: Drug: Pembrolizumab injection; Drug: Capecitabine tablets; Radiation: Local radiotherapy
- Standard of care (SOC) treated external cohort (Other): A standard of care treated external cohort with patients treated with pembrolizumab as postoperative treatment for localized TNBC without pCR after NAC, and with similar eligibility criteria will be registered in an ambispective way, allowing comparisons between the experimental arm and this external cohort. All the centres involved in the study will participate the registration of the needed information concerning this cohort.
  Interventions: Drug: Pembrolizumab injection; Radiation: Local radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab injection — On Day 1 of each cycle for a total of 9 cycles; intravenous (IV) infusion
  Other Names: KEYTRUDA®
Drug: Capecitabine tablets — 1250 mg/m² BID, on days 1-14 of each 21-day cycle; 8 cycles Dose reduction at 825 mg/m² BID during radiotherapy if indicated
  Other Names: Biogaran Capecitabine
  Arms: Experimental arm : Pembrolizumab and capecitabine
Radiation: Local radiotherapy — Local radiotherapy will be performed as per standard practice if indicated.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacity and safety of pembrolizumab and capecitabine on the invasive disease-free survival, in participants who have triple negative breast cancer (TNBC) with residual disease after neoadjuvant chemotherapy associated with pembrolizumab.

DETAILED DESCRIPTION:
We propose to evaluate the benefit in 2-year iDFS and safety of adding capecitabine to pembrolizumab in post-operative phase of pembrolizumab-containing treatment, in the subgroup of localized TNBC patients with residual disease.

An external cohort with patients treated with pembrolizumab as part of standard care after surgery, for localized TNBC without pCR after NAC, and with similar eligibility criteria, will be registered in an ambispective way, allowing comparisons between the experimental arm and this external cohort. All the centers involved in the study will participate in the registration of the needed information concerning this cohort.

ELIGIBILITY:
• CRITERIA FOR EXPERIMENTAL ARM :

Inclusion criteria (for experimental arm):

Patients eligible for this study must meet ALL of the following criteria:

1. Patient must have signed a written informed consent prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent;
2. Subject ≥18 years of age on day of signing informed consent form (ICF);
3. Histologically proven TNBC defined as follows:

   1. HER2 negativity (ASCO/CAP criteria)
   2. AND less than 10% of cells stained by immunohistochemistry (IHC) for ER and PgR;
4. TNBC patients previously treated by standard neoadjuvant chemotherapy with a minimum of 6 cycles of immunochemotherapy containing pembrolizumab, per standard of care (and pembrolizumab label) and anthracyclines and/or taxanes (with/without carboplatin). Other drugs may be acceptable following discussion with the sponsor (with the exclusion of capecitabine);
5. Complete resection of the breast tumor(s) (and of any invaded lymph node);
6. No complete pathological response, defined as RCB Class I, II or III (per local assessment);
7. Available representative formalin-fixed paraffin-embedded (FFPE) tumor block from surgery specimen with its histological report;
8. Eastern Cooperative Oncology Group (ECOG) Performance Status <2;
9. Adequate organ and bone marrow function. All screening lab tests should be performed within 28 days before inclusion;
10. Resolution to at least grade 1 of all acute toxicities from previous therapies including immune-related toxicity due to pembrolizumab, except alopecia and grade 2 immune-related endocrinopathies controlled by hormone replacement which are allowed;
11. Minimal/maximal period for prior treatments (i.e. minimal delay from last dose of prior treatment to C1D1): breast surgery (the wound must have healed prior to C1D1) ≥2 weeks (maximum 10 weeks); last pembrolizumab injection ≥3 weeks;
12. Women of child-bearing potential must have a negative serum pregnancy test within 7 days before C1D1;
13. Women of child-bearing potential and male patients must agree to use 1 effective form of contraception from the time of the negative pregnancy test up to 6 months after the last dose of study drugs;
14. Patient should be able and willing to comply with study visits and procedures as per protocol;
15. Patients must be affiliated to a Social Security System (or equivalent).

Non-inclusion criteria (for experimental arm):

Patients eligible for this study must not meet ANY of the following criteria:

1. Radiological or clinical evidence of metastatic disease documented by imaging or clinical examination performed during screening period;
2. Has received capecitabine or other ICI than pembrolizumab in the NAC regimen;
3. Has a known additional malignancy, excepted skin basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer or previously treated malignancy with no evidence of disease for ≥2 years;
4. Presents a contraindication to continue pembrolizumab treatment as per respective SmPC including known hypersensitivity;
5. Previous immune-related adverse event of any grade due to pembrolizumab that led to permanent discontinuation of pembrolizumab;
6. Presents a contraindication to capecitabine treatment as per SmPC (See EMA website for most recent edition of SmPC);
7. Complete DPD (Dihydropyrimidine Dehydrogenase) deficiency (a systematic screening of DPD deficiency must be performed);
8. Patient with active infection ;
9. Patients with history of uncontrolled or symptomatic cardiac disease ;
10. Patients having received brivudine within 4 weeks prior to inclusion;
11. Require the use of one of the following forbidden treatments during the study treatment period:

    * Any investigational anticancer therapy other than the protocol specified treatment;
    * Any concurrent chemotherapy, immunotherapy, biologic for cancer treatment, other than the ones stated in the protocol;
12. Pregnant women or women who are breast-feeding;
13. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons;
14. Persons deprived of their liberty or under protective custody or guardianship;
15. Participation in another therapeutic trial within the 30 days prior to randomization.

    * CRITERIA FOR STANDARD OF CARE TREATED EXTERNAL COHORT

Inclusion criteria (for standard of care treated external cohort) :

Patients eligible for this cohort must meet ALL of the following criteria:

1. Patient information prior to study entry and non-opposition to data collection
2. Subject ≥18 years of age ;
3. Histologically proven TNBC defined as follows:

   1. HER2 negativity (ASCO/CAP criteria)
   2. AND less than 10% of cells stained by immunohistochemistry (IHC) for ER and PgR;
4. TNBC patients previously treated by standard neoadjuvant chemotherapy with a minimum of 6 cycles of immunochemotherapy containing pembrolizumab, per standard of care (and pembrolizumab label) and anthracyclines and/or taxanes (with/without carboplatin). Other drugs may be acceptable following discussion with the sponsor (with the exclusion of capecitabine);
5. Complete resection of the breast tumor(s) (and of any invaded lymph node);
6. No complete pathological response, defined as RCB Class I, II or III (per local assessment);
7. Patient should have received at least one injection of pembrolizumab as post-surgery treatment (concomitantly or after radiotherapy).

Non-exclusion criteria (for standard of care treated external cohort) :

Patients eligible for this study must not meet ANY of the following criteria:

1. Radiological or clinical evidence of metastatic disease documented by imaging or clinical examination after surgery.
2. Has received capecitabine or other ICI than pembrolizumab in the NAC regimen;
3. Has a known additional malignancy, excepted skin basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer or previously treated malignancy with no evidence of disease for ≥2 years;
4. Any investigational anticancer therapy (chemotherapy, immunotherapy, biologic for cancer treatment) other than pembrolizumab only as adjuvant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
2-year Invasive Disease-free survival (iDFS) | 2 years
  Invasive disease free survival (iDFS) defined as time from randomization to the first of the following events: local, regional or distant recurrence, or second primary cancer (including contralateral) or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | From inclusion to death of any cause, up to 3.5 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Distant disease-free survival (DDFS) | Throughout study completion, up to 3.5 years.
  Distant disease-free survival (DDFS) is defined as the time from the date of inclusion to the date of distant relapse or death due to any cause, whichever occurs first.
Efficacy (iDFS, OS and DDFS) | Throughout study completion, up to 3.5 years.
  iDFS, OS and DDFS will also be compared to the external cohort of TNBC patients without pCR after NAC and treated with adjuvant pembrolizumab as part of standard of care after surgery .
Acute and late toxicity during the study | Throughout study completion, up to 3.5 years.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine LOIRAT, MD PhD, Principal Investigator — Institut Curie Paris; Jean-Yves PIERGA, MD, Principal Investigator — Institut Curie Paris
Locations (20):
- France (20):
  - CHU Amiens Picardie_Site Sud, Amiens
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHU Jean Minoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges-François Leclerc, Dijon
  - CHD Vendee, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut Curie, Paris
  - Clinique de La Croix du sud, Quint-Fonsegrives
  - Institut Godinot, Reims
  - Institut Curie, Saint-Cloud
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, IUCT Oncopole, Toulouse
  - CHU Bretonneau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.